CLINICAL TRIAL: NCT06768905
Title: IOMAB-ACT: A Phase Ib/II Multi-institutional Study of 131 I-Apamistamab Followed by CD19-Targeted CAR-T Cell Therapy for Patients With Relapsed or Refractory (R/R) Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of IOMAB-ACT Followed by CAR-T Cell Therapy for Patients Relapsed or Refractory (Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Actinium Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Farrukh Awan, Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-1091; SCCC-03424
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Non Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Safety run-in) (Experimental): 131I-Apamistamab dose will be given 5-7 days prior to a single infusion of CD-19 CAR-T cell therapy
  Interventions: Drug: Iomab-B; Drug: CAR-T cell
- Part B (cohort expansion) (Experimental): 131I-Apamistamab dose will be given 5-7 days prior to a single infusion of CAR-T cell therapy
  Interventions: Drug: Iomab-B; Drug: CAR-T cell

INTERVENTIONS:
Drug: Iomab-B — single 50 mCi dose of 131I-Apamistamab given prior to CAR-T cell infusion.
  Other Names: Iomab-ACT; 131I-Apamistamab
Drug: CAR-T cell — CAR-T cell therapy
  Other Names: CAR-T cell therapy

SUMMARY:
This study is being done to determine the safety, efficacy and tolerability of a single 50 mCi dose of 131I-Apamistamab given prior to CAR-T cell infusion in patients with Relapsed or refractory (R/R) Diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is an open-label single-cohort multi-institutional study of 131I-Apamistamab followed by CAR-T cell therapy for patients with (R/R) DLBCL. Patients will receive a 50 mCi single planned 131I-Apamistamab dose prior to CAR-T cell infusion for lymphodepleting conditioning. There will be a 6-patient safety run-in to assess safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diffuse large B-cell lymphoma (de novo or DLBCL transformed from an indolent lymphoma (follicular lymphoma, chronic lymphocytic leukemia [Richter syndrome]) or high-grade B-cell lymphoma (HGBL): ("DLBCL patients")

   * Defined as relapsed or refractory DLBCL or high-grade B-cell lymphoma (HGBL) following at least one or more prior chemoimmunotherapy regimen (with at least one course including an anthracycline and CD20-directed therapy) following diagnosis of de novo DLBCL/HGBL or DLBCL arising from indolent lymphoma and requiring further treatment and deemed to be candidates for standard of care CAR-T therapy. This includes patients with primary refractory disease (failure to achieve complete response (CR) to first-line therapy), relapsed disease within 12 months of first line chemoimmunotherapy or relapsed/refractory disease after 2 or more prior lines of systemic therapy.
   * Patients must have at least one FDG-avid (PET-avid) measurable lesion.
   * Relapsed or refractory disease must be confirmed with a repeat biopsy within the last 12 months.
   * For patients who have received treatment for confirmed relapsed or refractory disease otherwise meeting criteria 1.i.-1.iii. as above within 6 weeks of study enrollment, active disease does not need to be re-confirmed or present immediately prior to Screening 1 (Section 5.2) for the patient to be eligible for leukapheresis. However, detectable evidence of residual malignancy must be present at Screening 2 (Section 5.3) for the patient to be eligible for 131I-Apamistamab and CAR T-cell therapy.
2. Age ≥ 18 years of age
3. Creatinine clearance ≥50 mL/min as calculated by the Cockroft-Gault formula.
4. Total bilirubin ≤1.5x upper limit of normal , AST and ALT ≤3x upper limit of normal (ULN), unless liver dysfunction is thought to be related to underlying malignancy or secondary to Gilbert's disease in which case the direct bilirubin should be ≤3.0 mg/dL, and AST and ALT ≤5x ULN.
5. Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air or per institutional guidelines.
6. Thyroid function tests (TSH, FT4) ≤2x upper limit of normal (ULN)
7. Adequate bone marrow function meeting the following criteria as defined below, without requiring blood product or granulocyte-colony stimulating factor support in the 7 days prior to screening and start of 131I-Apamistamab treatment.

   1. Absolute neutrophil count ≥1.0k/µL,
   2. Platelets ≥50k/µL,
   3. Hemoglobin ≥8g/dL.
8. Performance status: ECOG performance status 0-2.
9. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, and/or abstinence) prior to study entry, and for the duration of study treatment, and for 30 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Ability to understand and the willingness to sign a written informed consent.
11. For patients undergoing bridging therapy after leukapheresis and prior to 131I-Apamistamab infusion a repeat PET/CT scan will be performed 10-14 days prior to the 131I-Apamistamab infusion. They will also be required to meet additional inclusion criteria as written within specific sections of the protocol within 10-14 days prior to the planned infusion of 131I-Apamistamab. This will be considered eligibility Screening 2 and will be approved by the Sponsor-Investigator.

Exclusion Criteria:

1. Pregnant or lactating patients.
2. Impaired cardiac function (LVEF <40%) as assessed by echocardiogram or MUGA scan.
3. Patients with active graft versus host disease following allogeneic hematopoietic cell transplantation requiring systemic T-cell suppressive therapy are ineligible.
4. Patients with active autoimmune disease requiring systemic T-cell suppressive therapy are ineligible.
5. Patients with the following cardiac conditions will be excluded:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure
   2. Myocardial infarction ≤6 months prior to enrollment
   3. Any history of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration.
6. Have current or prior positive test results for human immunodeficiency virus (HIV) or hepatitis B (HBV) or C (HCV), with the following exceptions:

   1. Patients who have positive HBV test results due to having been previously vaccinated against hepatitis B, as evidenced by negative hepatitis B surface antigen (HbsAg), negative anti- hepatitis B core protein (HBc) and positive antibody to the HbsAg (anti-HBs) are not excluded.
   2. Patients who have antibodies to HCV or who have hepatitis B core antibody, with undetectable viremia by PCR, and with adequate organ function as defined in the protocol, are not excluded.
7. Patients with uncontrolled systemic fungal, bacterial, viral, or other infections are ineligible.
8. Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of skin.
9. Patients with history or presence of clinically significant neurological disorders such as epilepsy, generalized seizure disorder, severe brain injuries are ineligible.
10. Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study.
11. Patients with circulating human anti-mouse antibodies (HAMA) to BC8
12. Patients with prior history of treatment with radiopharmaceuticals for any indication.
13. Patients with a history of external beam radiation therapy except for treatment of cutaneous lesions and localized prostate cancer.
14. Patients with QTcF >470mSec on EKG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (safety) -Part A (safety run-in) | Start of treatment up to 30 days post CAR T-cell infusion
  The number and percentage of patients with DLTs will be summarized for Part A using the DLT Analysis Set. The data analysis set will include all patients in Part A who received study medication and either experienced a DLT or completed at least 75% of the DLT period.
  Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.
Complete response (efficacy) -Part B (Cohort expansion) | Screening visit to Day 100 visit
  Measurement of effect (response and progression) will be conducted using a PET/CT scan which will report the Lugano criteria for response at screening 1 and 2 (if PET available), Day 30 +7 days, and Day 100 +/-7 days

SECONDARY OUTCOMES:
Severity of cytokine release syndrome (CRS) | within 100 days of CAR T-cell infusion
  Incidence and severity of CRS (all grades, as well as grade ≥3 CRS) following 131I-Apamistamab and CAR-T cell infusion in patients with R/R DLBCL will be collected.
  The number and percent of subjects developing versus not developing grade ≥3 neurologic toxicity following 131I-Apamistamab and CAR-T cell infusions will be summarized using the EAS. Efficacy Analysis Set (EAS): is defined as all patients in the SAS who have at least one post-baseline response assessment or discontinued the study due to disease progression (including death caused by disease progression).
Severity of immune effector cell-associated neurotoxicity (ICANS) | within 100 days of CAR T-cell infusion
  Neurologic toxicities (ICANS) will be graded by The American Society for Blood and Marrow Transplantation (ASBMT) Consensus Grading criteria for ICANS. The number and percent of subjects developing versus not developing grade ≥3 neurologic toxicity following 131I-Apamistamab and CAR-T cell infusions will be summarized using the EAS. Efficacy Analysis Set (EAS): is defined as all patients in the SAS who have at least one post-baseline response assessment or discontinued the study due to disease progression (including death caused by disease progression).

CONTACTS AND LOCATIONS:
Overall Officials: Farrukh Awan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided